CLINICAL TRIAL: NCT05196672
Title: Strategy Establishment of Promoting Sleep Quality and Quantity in Critically Ill Patients: The Effect and Mechanism of Guided-virtual-reality Autogenic Meditation
Brief Title: Effects and Mechanism of Guided Virtual Reality Autogenic Meditation on ICU Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the pandemic, is difficult to recruit the participants
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associated professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202104057
Record Dates: First submitted 2021-12-09; First posted 2022-01-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2022-01

CONDITIONS: Critical Illness; Sleep Quality
Keywords: intensive care unit; Sleep Disturbance; Virtual reality
MeSH Terms: conditions — Critical Illness; Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality (Experimental): Participants will receive virtual reality for 30 minutes before bedtime and then will be placed on an eye mask for a whole night's sleep for consecutive two days or until discharge from ICU. A total treatment dosage of 60 minutes is required.
  Interventions: Behavioral: Virtual reality and eye mask
- Eye masks (Experimental): Participants will receive eye masks during their sleep for consecutive two days or until discharge from ICU.
  Interventions: Behavioral: Virtual reality and eye mask
- Control group (No Intervention): The control group only receive routine care.

INTERVENTIONS:
Behavioral: Virtual reality and eye mask — Adults will receive a virtual reality program 30 min before bedtime and then be placed on an eye mask during their sleep for consecutive 2 nights of ICU stay.
  Arms: Eye masks; Virtual reality

SUMMARY:
Background: Sleep disturbance is a common complaint reported by critically ill patients, which may in turn prolong the length of intensive care unit (ICU) stay, and increase the risks of delirium and mortality. Environmental factors, such as noise and light exposures contribute to the development of sleep disturbances in ICU. Hypnotics is the most prescribed treatment for managing ICU sleep; however, it only improves light sleep but not deep sleep, and could not deal with sleep disturbances caused by noise or light exposure.

Purposes: To examine the effects of guided virtual reality autogenic meditation on sleep quality and quantity in critically ill adults as well as the possible mechanism through which they provide this alleviation. We hypothesize that critically ill adults undergoing guided virtual reality autogenic meditation (VR) will experience greater alleviations in sleep disturbances in comparison with participants in the eye masks and usual care control group (UC).

Methods: The three-year, single-blinded randomized controlled trial will employ a three-arm parallel-group design. A total of 120 critical ill adults will be randomly allocated to the VR, Eye masks, or UC groups in a 1:1:1 ratio (40 participants in each group). For the VR group, all participants will experience 30-min, voice-guided autogenic meditation through head-mounted display device at 10 pm for 2 nights (ICU day 2 to day 4). For the Eye masks group, participants will wear eye mask from 10 pm to 7 am for 3 days. For the UC group, they will receive sleep promotion strategies, including reduced light exposure at night, decreased noise, and cluster nursing care during the study period. Primary outcomes are sleep parameters measured by the Chinese version of Richards-Campbell Sleep Questionnaire, Chinese version of Pittsburgh sleep quality index, and fitbit with one-lead electroencephalography sensor. Secondary outcomes consist of delirium, moods, and quality of life assessed using the Confusion Assessment Method for the Intensive Care Unit, visual analogue scale for anxiety, pain, stress, EuroQoL-5D, and cognitive function respectively. Measurement time points are the first day of ICU admission, pre-and post-treatment, and the day of 30 and 180 days after ICU discharge. A generalized estimating equation will be used to test research hypotheses.

DETAILED DESCRIPTION:
Sleep disturbance has affected up to 59% of patients who are admitted into intensive care units (ICUs). Such disturbance has been associated with prolonged ICU length of stay, the occurrence of delirium, increased medical costs. The risk factors related to poor sleep in ICU patients include bright light, artificial/augmented sound, postoperative pain, prior illness status, higher intensity of care, and equipment applications.

To date, pharmacological and nonpharmacological therapies have been widely used to relieve poor sleep in ICU. Sedative-hypnotic is the most prescribed treatment for critically ill patients with sleep problems. However, related adverse events reduce their usefulness.

According to the 2018 PADIS guideline of the Society of Critical Care Medicine, sleep disturbance has been listed as one of the critical symptoms that must be recognized in a critically clinical setting. Recently, technology-assisted interventions have been increasingly integrated into critical care. Virtual reality (VR) mediation is a promising technology for free from time and space that provides various contents or games to users. To achieve the goal of precision health, more researchers and health care providers have incorporated high technology into medical and nursing care systems. Thus far, only one randomized controlled trial involving 52 ICU patients investigated the effect of VR meditation (natural scenes and sounds) on poor sleep quality and found that the program significantly decreased wake after sleep onset and increased deep sleep time. Therefore, we aim to develop a new VR-assisted program and to examine its effects on sleep quality and quantity of adults requiring intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years and above.
* Clear consciousness and able to communicate with Chinese or Mandarin.
* Expect to stay in ICU for more than 72 hrs

Exclusion Criteria:

* The use of invasive mechanical ventilation.
* Having visual or hearing difficulty
* Having a medical history of sleep disorder, cognition impairment, psychiatric disorders, or seizures.
* Having sedation use
* Having APACHE II over 25

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Changes in subjective sleep quality from 1st day and 2th day after ICU admission | The 1st, and 2th night after ICU admission
  Subjective sleep quality in ICU is assessed by Richards-Campbell Sleep Questionnaire(RCSQ). The mean of total score is 0-100. The higher score means the better sleep quality.
Change of subjective sleep quality before ICU admission and 30 and 180 days days after ICU discharge | The first day of ICU admission, 30 and 180 days days after ICU discharge
  Subjective sleep quality is assessed by Pittsburgh Sleep Quality. Index(PSQI). The total score is 0-21. The higher score means the worse sleep quality.
Changes in subjective sleep quality from 1st day and 2th day after ICU admission | The first night and 2th night of ICU stay
  Objective sleep quality in ICU is measured by fitbit

SECONDARY OUTCOMES:
Change of quality of life from the first day of ICU admission, 30 and 180 days after ICU discharge | The 1st day of ICU admission, 30 and 180 days days after ICU discharge
  Quality of life is assessed by EuroQol- 5 Dimension(ED-5D). The total score is 0-100.The higher score means the better quality of life.
Delirium occurrence | The 1st to 3th days of ICU admission
  Delirium is assessed by Confusion Assessment Method for the ICU (CAM-ICU).
Change of heart rate variability | The 1st to 2th days of ICU admission
  Heart rate variability is measured by portable ECG recorder and analyzer.
Change from baseline on anxiety | The 1day (date of enrollment)and up to 30 and 180 days
  Anxiety is assessed by Visual Analog Scale (VAS) anxiety scoring.The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain(score of 10) .The higher score means the very anxiety.
Electroencephalography | The first day to 3th day of ICU admission
  Electroencephalography is measured by Neurosky mindwave mobile 2
Change of stress | The first day of ICU admission, 30 and 180 days after ICU discharge
  Stress is assessed by Visual Analog Scale(VAS) stress scoring.The scale is most commonly anchored by "no stress" (score of 0) and "very stressful(score of 10) .The higher score means the very stressful.
Change of pain | The first day of ICU admission, 30 and 180 days days after ICU discharge
  Pain is assessed by Visual Analog Scale(VAS) pain scoring.The scale is most commonly anchored by "no pain" (score of 0) and "very painful(score of 10) .The higher score means the very painful.
Change of cognitive function | The 30 and 180 days after ICU discharge
  Cognitive function is assessed by MoCA. The total scales is 30. The scale is more than 26 means the patients do not have cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, PhD, Study Director — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No